CLINICAL TRIAL: NCT01195298
Title: Phase II Clinical Study of Bevacizumab in Combination With Capecitabine as First-line Treatment in Elderly Patients With Metastatic Breast Cancer
Brief Title: Bevacizumab and Capecitabine in Treatment of Elderly Patients With Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: South Eastern European Research Oncology Group (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Prof. dr. sc. Eduard Vrdoljak, Clinical Hospitl Split, Center of oncology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML22373
Record Dates: First submitted 2010-08-26; First posted 2010-09-06 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-08

CONDITIONS: Breast Cancer; Metastasis
Keywords: metastatic breast cancer; elderly patients; chemoimmunotherapy; Triple negative metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Capecitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Capecitabine and Bevacizumab — Drugs will be administered in 3-week cycles as follows:
  * Bevacizumab 15mg/kg via i.v. infusion on day 1
  * Capecitabine 1000 mg/m2 tablets twice-daily, on days 1 through 14.
  Other Names: Bevacizumab (Avastin ); Capecitabine (Xeloda)

SUMMARY:
This is an open-label, single-arm, multicenter study of capecitabine and bevacizumab administered as first-line treatment of previously untreated elderly patients, older than 70 years, with metastatic or locally recurrent breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained prior to initiation of any study specific procedures and treatment as confirmation of the patient's awareness and willingness to comply with the Protocol code: ML22373 Protocol SEEROG: version 1.2. Date: October 15, 2009 3 study requirements;
* Age ≥70 years;
* Pathologically confirmed and documented metastatic breast cancer or locally recurrent breast cancer not amenable to curative treatment. Complete radiology and tumor measurement workup must be completed within 4 weeks prior to first study treatment;
* Measurable disease according to RECIST criteria;
* HER2 negative disease;
* No prior treatment for metastatic or locally recurrent disease;
* Prior radiotherapy is allowed if delivered at least 2 weeks before enrolment in the study and for the relief of metastatic bone pain, and provided that no more than 30% of marrow bearing bone was irradiated and that target lesions were not included in the radiotherapy field;
* Not suitable for aggressive chemotherapy regimen in the opinion of the investigator;
* Performance status ECOG 0 - 2.

Exclusion Criteria:

* Any prior neoadjuvant or adjuvant treatment with anthracyclines completed less than 6 months prior to enrolment. The maximum cumulative dose received must not have exceeded 360 mg/m2 for doxorubicin or 720 mg/m2 for epirubicin. Prior anti-epidermal growth factor therapy is allowed;
* Concurrent hormonal therapy; however previous hormonal therapy is allowed for adjuvant, locally recurrent, or metastatic breast cancer if completed within ≥1 months prior to enrolment;
* History or clinical evidence of brain metastases. If there is any clinical suspicion of brain metastasis, a computerized tomography (CT) scan or magnetic resonance imaging (MRI) of the brain must be conducted within 4 weeks prior to enrolment;
* Other malignancy (including primary brain tumors) within the Protocol code: ML22373 Protocol SEEROG: version 1.2. Date: October 15, 2009 4 last 5 years, which could affect the diagnosis or assessment of breast cancer, except for adequately treated carcinoma in situ of the cervix, squamous carcinoma of the skin, or adequately controlled limited basal cell skin cancer;
* Life expectancy < 12 weeks;
* Any of the following abnormal values:

  * Inadequate bone marrow function: hemoglobin (Hb) < 8.0 g/dL, absolute neutrophil count (ANC) < 1.5 x 109/L, or platelet count < 100 x 109/L;
  * Inadequate liver function: AST/SGOT or ALT/SGPT > 2.5 x upper limit of normal (ULN) or > 5 x ULN in patients with liver metastases), serum alkaline phosphatase > 2.5 ULN or > 5 x ULN in patients with liver metastases, or > 10 x ULN in patients with bone metastases or total bilirubin > 2 x ULN;
  * Moderate or severe renal impairment: creatinine clearance ≤50 mL/min (calculated according to the cockcroft and Gault formula; see Appendix 1), or serum creatinine > 1.5 x ULN;
* Chronic daily treatment with aspirin (> 325 mg/day) or clopidogrel (> 75 mg / day);
* Chronic daily treatment with corticosteroids (dose of > 10 mg/day methylprednisolone equivalent) (excluding inhaled steroids);
* Requirement for concurrent use of the antiviral agents sorivudine or brivudine;
* Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to enrolment, or anticipation of the need for major surgery during the course of the study treatment;
* Minor surgical procedures, within 24 hours prior to enrolment;
* Current or recent (within the 30 days prior to starting study treatment) treatment with another investigational drug or participation in another investigational study.
* Uncontrolled hypertension (systolic > 150 mm Hg and/or diastolic > 100 mm Hg) or clinically significant (i.e. active) cardiovascular disease, including:
* Cerebrovascular accident/stroke (≤ 6 months prior to enrolment)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
Time to treatment progression | average 5 years
  followed until death

SECONDARY OUTCOMES:
overall response rate in patients with measurable disease at baseline | average 5 years
safety and tolerability | average 5 years
Clinical benefit (complete response, partial response and stable disease) in patients with measurable disease at baseline | average 5 years
progression-free survival | average 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vrdoljak, PhD MD, Principal Investigator — Clinical Hospital Split, Center of oncology, Croatia; Damir Vrbanec, PhD MD, Principal Investigator — Clinical Hospital Zagreb, Croatia; Katarina Petrakova, MD, Principal Investigator — Masaryk Memorial Cancer Institue, Brno, Czech Republic; Gyorgy Bodoky, PhD MD, Principal Investigator — FOVAROSI SZENT LASZLO KORHAZ-RENDELOINTEZET, ONKOLOGIAI OSZTALY, Budapest, Hungary; Tamas Pinter, MD, Principal Investigator — Petz, Aladar Korhaz, Onkoradiologiai Osztaly, Gyor, Hungary; Vladimir Todorović, MD, Principal Investigator — Oncology clinic, Clinical Center of Montenegro; Marek Wojtukiewicz, PhD MD, Principal Investigator — Department of Oncology Medical University, Bialystok, Poland; Tadeusz Pienkowski, PhD MD, Principal Investigator — Cancer Centre and Institute of Oncology Warsaw; Daniela Grecea, MD, Principal Investigator — "Prof Dr. I Chiricuta" Cluj Napoca Oncology Institute - Breast Cancer Center, Cluj Napoca, Romania
Locations (1):
- Clinical Hospital Split, Center of oncology, Split, Croatia